CLINICAL TRIAL: NCT02178228
Title: Prospective Assessment of Anastomotic Leak
Brief Title: Observational Analysis of the Cause of Leaks When Bowel is Cut and Reconnected
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: ECRI Institute (Unknown); Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: GCO 09-2235
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Anastomotic Leaks
Keywords: Anastomotic Leaks; Bowel Resection; Postoperative Complication
MeSH Terms: conditions — Anastomotic Leak; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects over age 18: Subjects undergoing non-emergent small bowel or large bowel surgery and reconnection of bowel that are over the age of 18
- Subjects age 15-17: Subjects undergoing non-emergent small bowel or large bowel surgery and reconnection of bowel that are age 15-17 with one permission of one parent.

SUMMARY:
The purpose of this study is to identify the cause of leaks that sometimes occur after a section of the bowel is removed and reconnected. Certain staplers from the operating room will be collected and sent to a third party (ECRI Institute) to be examined for defects. The patient's charts will be analyzed for medical issues that may contribute to leaks after surgery.

DETAILED DESCRIPTION:
The objective of this study is to identify peri-operative factors that contribute to leaks after a portion of the bowel has been cut and reconnected. Most specifically, the role of staplers in this reconnection of the bowels will be evaluated. The research will take place at Icahn School of Medicine where there is an extremely high volume of operations involving small bowel and large bowel being cut and reconnected. Patients will be recruited based on inclusion and exclusion criteria and 500 subjects are expected to be enrolled in the study. The surgery will be performed in a standard fashion as indicated by diagnosis, location of disease, patient condition, and surgeon preference. No changes to the surgical procedure will be mandated by the research protocol. This is purely an observational study with no changes to the standard of care. The patients will be followed throughout the course of the their hospital stay for the scheduled surgery up to one week and one month after the procedure to gather laboratory data and any complications incurred due to the surgery. No patient specimen will be stored. The staplers used in the procedure will be collected, stored in sterile plastic container, information about the staplers will be recorded, and then discarded after 30 days in the usual manner that the operating room staff employs to discard the staplers. Subjects lost to follow-up after the procedure will be withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be scheduled for non-emergent small or large bowel surgery and reconnection of bowel at Icahn School of Medicine at Mount Sinai
* Subjects must be able and willing to provide informed consent
* Subjects must be 18 years or above OR 15-17 with permission of one parent
* English and Spanish speaking patients will be included in this study

Exclusion Criteria:

* Subject who are less than 15 years of age
* Subject who are scheduled for emergent surgery, precluding the capacity to give informed consent
* Subjects who are diagnosed with obstructed or perforated colon cancer

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are scheduled to have a small or large bowel surgery and reconnection of bowel will be selected from the operating room schedule at Icahn School of Medicine at Mount Sinai.
Sampling Method: Non-Probability Sample
Enrollment: 1077 (Actual)
Dates: Start 2013-10; Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
All cause bowel leaks after surgery | one week post-operation
All cause bowel leaks after surgery | one month post-operation

SECONDARY OUTCOMES:
Reoperation | 1 year post operation
Sepsis | 1 year post operation
Length of hospital stay | 1 year post operation
Mortality | 1 year post operation

CONTACTS AND LOCATIONS:
Overall Officials: Celia Divino, M.D. FACS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States